CLINICAL TRIAL: NCT01410253
Title: Evaluation of the Effects of Different Physical Therapy on Cardiac Rehabilitation in Post Operatory Period of Coronary Artery Bypass Graft: Randomized Clinical Trial.
Brief Title: Effects of Cardiac Rehabilitation on Postoperatory of Coronary Artery Bypass Graft.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Maurice Zanini, Msc., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GPPG090650
Record Dates: First submitted 2011-05-10; First posted 2011-08-05 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Complication of CABG
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental)
  Interventions: Other: Combination of four techniques of physiotherapy
- Group 2 (Experimental)
  Interventions: Other: Combination of three techniques of physiotherapy
- Group 3 (Experimental)
  Interventions: Other: Combination of two techniques of physiotherapy
- Group 4 (Placebo Comparator)
  Interventions: Other: standard therapy

INTERVENTIONS:
Other: Combination of four techniques of physiotherapy — The patients receive conventional physiotherapy, expiratory positive airway pressure, inspiratory muscle training and physical exercise. Twice daily for seven days
  Arms: Group 1
Other: Combination of three techniques of physiotherapy — Patients receive conventional physiotherapy, expiratory positive airway pressure and physical exercise. Twice daily for seven days
  Arms: Group 2
Other: Combination of two techniques of physiotherapy — Patients receive conventional physiotherapy,expiratory positive airway pressure respiratory muscle training. Twice daily for seven days
  Arms: Group 3
Other: standard therapy — Patients receive conventional physiotherapy and expiratory positive airway pressure. Twice daily for seven days
  Arms: Group 4

SUMMARY:
Randomized Clinical Trial to evaluate the use of different techniques of physical therapy on recovery of functional capacity, pulmonary function and respiratory muscle strength in the period of hospital stay after coronary artery bypass graft.

ELIGIBILITY:
Inclusion Criteria:

-Patients are recruited from the waiting list for a first CABG intervention at the Porto Alegre Clinical Hospital.

Exclusion Criteria:

* chronic renal failure,
* unstable angina,
* moderate or severe valve disease,
* complex cardiac arrhythmia,
* stroke,
* inability to exercise the lower limbs,
* subjects with forced expiratory volume in 1 second less than 70% of predicted

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2015-11 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
submaximal functional capacity | Change from Baseline in functional capacity at seven days and thirty days after surgery
  functional capacity evaluated by six-minute walk test

SECONDARY OUTCOMES:
capacity functional | evaluated 40 days after surgery
  cardiopulmonary exercise testing ( VO2)
respiratory muscle strength | Change from Baseline in respiratory muscle strength at seven days and thirty days after surgery
  Both PImax and PEmax were obtained using a pressure transducer
lung function | Change from Baseline in lung function at seven days and thirty days after surgery
  assessed by spirometry (FVC and FEV1)

CONTACTS AND LOCATIONS:
Locations (1):
- Porto Alegre Clinical Hospital, Porto Alegre, Rio Grande do Sul, Brazil